CLINICAL TRIAL: NCT06389461
Title: The Efficacy of the 4th Ventricular Compression Technique on Anxiety in Students: RCT
Brief Title: 4th Ventricular Compression Technique on Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OST1_012
Record Dates: First submitted 2024-04-16; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Anxiety; College Students; CV4; Osteopathic treatment
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4th Ventricular Compression Technique (Experimental): The technique was preformed by the investigator during 5 minutes.
  Interventions: Other: 4th Ventricular Compression Technique
- "Sham" Therapy (Placebo Comparator): The technique was preformed by the investigator during 5 minutes.
  Interventions: Other: "Sham" Therapy

INTERVENTIONS:
Other: 4th Ventricular Compression Technique — The investigator who applied the technique stood on top of the headboard of the table, with feet flat on the floor, at an appropriate level in relation to the volunteer's headboard.
  The investigator joins hands in a cupping position, with the pads of the 1st fingers forming a triangle. The pads of the 1st fingers make contact with the spinous processes of the 2nd and 3rd cervical vertebrae. The thenar eminences make contact with the occipital squama, avoiding contact with the occipito-mastoid sutures during 5 minutes.
  A second Investigator was sitting on a chair, placed on the opposite side of the head of the table with a stopwatch in his dominant hand, in order to time the application time of each technique.
  Arms: 4th Ventricular Compression Technique
Other: "Sham" Therapy — The investigator who applied the technique stood on top of the headboard of the table, with feet flat on the floor, at an appropriate level in relation to the volunteer's headboard.
  The investigator places hands on the patient's shoulders during 5 minutes. A second Investigator was sitting on a chair, placed on the opposite side of the head of the table with a stopwatch in his dominant hand, in order to time the application time of each technique.
  Arms: "Sham" Therapy

SUMMARY:
Determinate the effects of the technique of 4th ventricle in college students with anxiety, applying the technique one time per week during three weeks.

DETAILED DESCRIPTION:
The anxiety is a warning sign that makes it possible for the individual to defend themselves and protect themselves from threats. This is considered a natural and necessary reaction for self-preservation. However, when it appears persistently, exaggeratedly or disproportionately in relation to a stimulus, the following are considered: pathological anxiety.

The compression of the fourth ventricle (CV4) is one of the most well-known procedures in the practice of cranial manipulation. It is also one of the most clinically tested techniques and has been postulated to be associated with decreased sympathetic tone.

Therefore, this was the chosen technique, as it significantly affects the relaxation of the SNS tonus and, thereafter, anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 25 years old;
* Be a college/university student;
* Not have knowledge of the technique used;
* Achieve a 20 plus score on the State-Trait Anxiety Inventory questionnaire.

Exclusion Criteria:

* Use of pharmacological therapy for psychological disorders;
* Presence of conditions that prevent or contraindicate the technique, including tumors, fractures, dislocations, vertebrobasilar insufficiency, bone diseases, neurological diseases, fever, skin diseases, cardiovascular diseases, psychiatric diseases, increased intracranial pressure.
* Surgeries or traumas in the specific areas of the technique;
* Pregnancy;
* Osteopathic treatments or other manual therapies aimed at reducing anxiety;
* Evident postural alteration or deformity of the thoracic cage.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-16 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in anxiety levels through the STAI (The State-Trait Anxiety Inventory) questionnaire score on the 1st and last intervention. | One week after the last intervention
  The participants were submitted to a evaluation 1 week prior the 1st and 1 week after the last intervention. The corresponding questionnaires were sent to the researchers so that they could record the information. Quoted with a min. of 20 points and a max. of 80 - higher the score worst level of anxiety.

SECONDARY OUTCOMES:
Change from baseline in thoraco-abdominal perimetry on the 1st and last intervention | Immediately after last intervention
  The participants were submitted to a evaluation/ measurement in the 1st and last intervention. The corresponding results were registered by the researchers so that they could record the information.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Natália, Principal Investigator — Escola Superior da Saúde do Porto
Locations (1):
- Escola Superior da Saúde do Porto, Porto, Portugal

REFERENCES:
- Available data/document: Castilloa, A. R. G. L., Recondob, R., Asbahrc, F. R. & Manfrod, G. G. (2000). — https://doi.org/10.1590/S1516-44462000000600006 — Transtornos de ansiedade. Revista Brasileira de Psiquiatria. 22(2), 20-23.
- Available data/document: Abenavoli, A., Badi, F., Barbieri, M., Bianchi, M., Biglione, G., Dealessi, C., Grandini, M., Lavazza, C., Mapelli, L., Milano, V., Monti, L., Seppia, S., Tresoldi, M. & Maggiani, A. (2020). — http://doi.org/10.1016/j.jbmt.2020.07.017 — Cranial osteopathic treatment and stress-related effects on autonomic nervous system measured by salivary markers: A pilot study. Journal of Bodywork and Movement Therapies. 24(4), 215-221.